CLINICAL TRIAL: NCT01763788
Title: An Open-Label, Multicenter, Phase 1b/2 Study to Evaluate Necitumumab in Combination With Gemcitabine and Cisplatin in the First-Line Treatment of Patients With Advanced (Stage IV) Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Necitumumab in the First-Line Treatment of Stage IV Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14461; I4X-JE-JFCM (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2018-12

CONDITIONS: Squamous Non-small Cell Lung Cancer
MeSH Terms: interventions — necitumumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Necitumumab + Gem and Cis (Experimental): Phase 1b Dose Escalation: Necitumumab 800 milligram (mg) on Days 1 and 8 of every 21 day cycle, administered as an intravenous (IV) infusion. Gemcitabine (Gem) dose escalation of 1000 or 1250 milligram per square meter (mg/m^2) on Days 1 and 8 of every 21 day cycle, administered as an IV infusion for a maximum of 4 cycles. Cisplatin (Cis) 75 mg/m^2 on Day 1 of every 21 day cycle, administered as an IV infusion for a maximum of 4 cycles.
  Phase 2 Randomized: Necitumumab 800 mg on Days 1 and 8 of every 21 day cycle, administered as an IV infusion. Gemcitabine at fixed dose determined in Phase 1b (1000 or 1250 mg/m^2) on Days 1 and 8 of every 21 day cycle, administered as an IV infusion for a maximum of 4 cycles. Cisplatin 75 mg/m^2 on Day 1 of every 21 day cycle, administered as an IV infusion for a maximum of 4 cycles.
  Interventions: Drug: Necitumumab; Drug: Gemcitabine; Drug: Cisplatin
- Gemcitabine + Cisplatin (Active Comparator): Phase 2 Randomized: Gemcitabine at fixed dose determined in Phase 1b (1000 to 1250 mg/m^2) on Day 1 and Day 8 of every 21 day cycle,administered as an IV infusion over approximately 30 minutes for a maximum of 4 cycles. Cisplatin 75 mg/m^2 on Day 1 of every 21 day cycle, administered as an IV infusion over approximately 120 minutes for a maximum of 4 cycles .
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Necitumumab — Administered IV
  Other Names: IMC-11F8; LY3012211
  Arms: Necitumumab + Gem and Cis
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
Drug: Cisplatin — Administered IV

SUMMARY:
The purpose of the Phase 1b portion of the study is to investigate how the body tolerates necitumumab, in combination with gemcitabine and cisplatin chemotherapy as first line treatment in participants with Stage IV squamous NSCLC and to determine the recommended dose for the subsequent Phase 2 portion of the study.

The purpose of the Phase 2 portion of the study is to evaluate the efficacy of necitumumab in combination with gemcitabine and cisplatin chemotherapy in participants with Stage IV squamous NSCLC in a first-line setting.

ELIGIBILITY:
Inclusion Criteria:

* Squamous Non-Small Cell Lung Cancer Disease (NSCLC)
* Clinical Stage IV NSCLC
* Measurable or nonmeasurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* No prior systematic chemotherapy, targeted therapy, surgery and chest radiotherapy
* Ha resolution to Grade less than or equal to (≤) 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0, of all clinically significant toxic effects of prior therapy for other than NSCLC
* Adequate-organ function defined as:
* Total bilirubin ≤1.5 x the upper limit of normal value (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Serum creatinine ≤ 1.2 x ULN or calculated creatinine clearance (CrCL)>50 milliliter per minute (mL/min) (per the Cockcroft Gault formula or equivalent and/or 24-hour urine collection)
* Absolute neutrophil count (ANC) greater than or equal to ≥1.5 x 10^3/μL(microliter)
* Hemoglobin ≥10.0 g/dL(gram per deciliter)
* Platelets ≥100 x 10^3/μL
* At least 20 years of age
* Estimated life expectancy of at least 12 weeks
* A formalin-fixed, paraffin-embedded tumor tissue block or a minimum of 5 unstained slides of tumor sample prior to randomization for the evaluation of epidermal growth factor receptor (EGFR) protein expression (IHC).
* If women: surgically sterile, postmenopausal, or compliant with a highly effective contraceptive method (failure rate <1%) during and for 6 months after the treatment period (oral hormonal contraception alone is not considered highly effective and must be used in combination with a barrier method). If men: surgically sterile or compliant with a highly effective contraceptive regimen during and for 6 months after the treatment period.
* Has provided signed informed consent

Exclusion Criteria:

* Has enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device
* Participant has undergone major surgery within 28 days prior to enrollment or have planned major surgery, subcutaneous venous access device placement within 7 days prior to enrollment Phase 1b) or randomization (Phase 2).
* Has undergone any prior radiation therapy, except for Gamma Knife radiation and palliative radiation treatment at least 14 days have elapsed from last radiation treatment prior to enrollment (Phase 1b) or randomization (Phase 2)
* Has brain metastases that are symptomatic or require surgery, medication and radiotherapy except for stereotactic irradiation
* Has superior vena cava syndrome
* Has clinically relevant coronary artery disease or uncontrolled congestive - heart failure
* Participant has uncontrolled hypertension defined as systolic blood pressure ≥150 mmHg or diastolic blood pressure ≥90 mmHg despite standard medical management.
* Has diabetes requiring insulin
* Has an angina or has experienced myocardial infarction within 6 months prior to enrollment (Phase 1b) or randomization (Phase 2)
* Has an Acquired Immunodeficiency Syndrome (AIDS)-related illness or have evidence of or test positive test results for human immunodeficiency virus (HIV)
* Has evidence of or test positive test results for hepatitis B, or hepatitis C virus antibodies
* Has a known allergy and history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab, or any other contraindication to one of the administered treatments
* Has significant third-space fluid retention requiring drainage
* Has history of interstitial pneumonitis
* Has an ongoing or active infection
* Has a history of significant neurological or psychiatric disorders
* Has a Grade 2 peripheral neuropathy
* Pregnant (confirmed within 7 days prior to enrollment [Phase 1b] or randomization [Phase 2]), or breastfeeding
* Has known history of drug abuse
* Assessed as inadequate for the study by the investigator or sub investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (20):
- Japan (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kōtoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wakayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Watanabe S, Yoshioka H, Sakai H, Hotta K, Takenoyama M, Yamada K, Sugawara S, Takiguchi Y, Hosomi Y, Tomii K, Niho S, Yamamoto N, Nishio M, Ohe Y, Kato T, Takahashi T, Kamada A, Suzukawa K, Omori Y, Enatsu S, Nakagawa K, Tamura T. Necitumumab plus gemcitabine and cisplatin versus gemcitabine and cisplatin alone as first-line treatment for stage IV squamous non-small cell lung cancer: A phase 1b and randomized, open-label, multicenter, phase 2 trial in Japan. Lung Cancer. 2019 Mar;129:55-62. doi: 10.1016/j.lungcan.2019.01.005. Epub 2019 Jan 16. PMID 30797492

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died from any cause and participants who were alive and on study (but off treatment) at study conclusion.
Groups:
- Phase 1b: Cohort 1: Gemcitabine at a dose of 1000 mg/m^2 (milligrams per square meter) was administered over approximately 30 minutes intravenously (IV) on Days 1 and 8 of each cycle for a maximum of 4 cycles.
  Cisplatin at a dose of 75 mg/m^2 was administered over approximately 120 minutes IV on Day 1 for a maximum of 4 cycles.
  Necitumumab at a dose of 800 mg was administered over approximately 50 minutes intravenously IV on Days 1 and 8 of each 3-week cycle.
- Phase 1b: Cohort 2; Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab): Gemcitabine at a dose of 1250 mg/m^2 was administered over approximately 30 minutes IV on Days 1 and 8 of each cycle for a maximum of 4 cycles.
  Cisplatin at a dose of 75 mg/m^2 was administered over approximately 120 minutes IV on Day 1 for a maximum of 4 cycles.
  Necitumumab at a dose of 800 mg was administered over approximately 50 minutes intravenously IV on Days 1 and 8 of each 3-week cycle.
- Phase 2: GC (Gemcitabine, Cisplatin): Gemcitabine at a dose of 1250 mg/m^2 was administered over approximately 30 minutes IV on Days 1 and 8 of each cycle for a maximum of 4 cycles.
  Cisplatin at a dose of 75 mg/m^2 was administered over approximately 120 minutes IV on Day 1 for a maximum of 4 cycles.
Period: Overall Study
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2 | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Started | 3 | 6 | 91 | 92
Received at Least 1dose of Study Drug | 3 | 6 | 90 | 91
Completed | 3 | 6 | 90 | 92
Not Completed | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Phase 1b: Cohort 1: Gemcitabine at a dose of 1000 mg/m^2 was administered over approximately 30 minutes IV on Days 1 and 8 of each cycle for a maximum of 4 cycles.
  Cisplatin at a dose of 75 mg/m^2 was administered over approximately 120 minutes IV on Day 1 for a maximum of 4 cycles.
  Necitumumab at a dose of 800 mg was administered over approximately 50 minutes intravenously IV on Days 1 and 8 of each 3-week cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2 | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin) | Total
Number analyzed (Participants) | 3 | 6 | 90 | 91 | 190
Age, Continuous [Median (Full Range); unit: years] | 71.0 [70 to 73] | 66.0 [59 to 74] | 66.5 [35 to 78] | 65.0 [31 to 77] | 66.0 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 11 | 10 | 22
  Male | 3 | 5 | 79 | 81 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 90 | 89 | 188
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following events graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, when the event occurred within 21 days from Day 1 in Cycle 1 and was considered to be definitely or probably related to necitumumab and/or gemcitabine-cisplatin chemotherapy: Grade 4 neutropenia ≥ 7 days, Grade ≥ 3 febrile neutropenia except for transient febrile neutropenia (Grade 3 neutropenia with fever ≥ 38.5 degrees Celsius (°C) for ≤ 24 hours), Grade 3 thrombocytopenia requiring platelet substitution, Grade 4 thrombocytopenia, ≥Grade 3 nonhematologic toxicity (excluding nausea, vomiting, arthralgia, myalgia, asthenia, fatigue, diarrhea, constipation, anorexia), any toxicity leading to the omission of necitumumab on Day 8 or 15 (for participants for whom necitumumab was delayed from Days 8 to 15) during the Cycle 1.
Time Frame: Day 1 to Day 21 in Cycle 1 (Up To 21 days)
Population: All enrolled participants who received at least one dose of study drug during study Phase 1b.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Phase 2: Overall Survival (OS)
Description: OS defined as the time from the date of randomization to the date of death due to any cause. Participants who are alive at the time of study completion or are lost to follow-up will be censored at the time they were last known to be alive.
Time Frame: From Date of Randomization until Death Due to Any Cause (Up To 39 Months)
Population: All randomized participants who received at least one dose of study drug during study Phase 2. Censored participants in the GC+N Arm = 27 and in the GC Arm = 17.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 90 | 91
Months | 14.92 [13.37 to 18.17] | 10.84 [8.90 to 14.39]
Statistical Analysis 1: Comparison: Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) vs Phase 2: GC (Gemcitabine, Cisplatin); Test type: Superiority; p = 0.0161, Stratified Log Rank; Stratified Hazard Ratio = 0.656, 95% CI 2-sided [0.465 to 0.926]

3. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS defined as time from date of randomization until first radiographic documentation of measured progressive disease(PD) defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. PD was at least 20% increase in sum of diameters of target lesions with reference being smallest sum on study and an absolute increase of at least 5 mm,or unequivocal progression of non-target lesions,or 1 or more new lesions.If participant does not have complete baseline disease assessment,PFS time censored at date of randomization,regardless of whether or not objectively determined disease progression or death observed for participant.If participant was not known to have died or have objective progression as of data inclusion cutoff date for analysis,the PFS time censored at last adequate tumor assessment date.The use of new anticancer therapy prior to occurrence of PD resulted in censoring at the date of last radiographic assessment prior to initiation of new therapy.
Time Frame: From Date of Randomization to Measured Progressive Disease or Death Due to Any Cause (Up To 39 Months)
Population: All randomized participants who received at least one dose of study during study Phase 2. Censored participants in the GC+N Arm = 6 and in the GC Arm = 10.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 90 | 91
Months | 4.21 [4.14 to 4.27] | 4.01 [3.52 to 4.17]

4. Secondary Outcome: Phase 1b: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response or Partial Response (Objective Tumor Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of nontarget lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Measured Progressive Disease (Up To 39 Months)
Population: All randomized participants who received at least one dose of study drug during study Phase 1b.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
percentage of participants | 0.0 [0.0 to 0.0] | 83.3 [53.5 to 100.0]

5. Secondary Outcome: Phase 2: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete Response or Partial Response (Objective Tumor Response Rate [ORR])
Description: as for outcome 4
Time Frame: Baseline to Measured Progressive Disease (Up To 39 Months)
Population: All randomized participants who received at least one dose of study drug during study Phase 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 90 | 91
percentage of participants | 51.1 [40.8 to 61.4] | 20.9 [12.5 to 29.2]

6. Secondary Outcome: Phase 2: Time to Treatment Failure (TTF)
Description: TTF was time from the date of randomization until the date of the first observation of radiographically documented progressive disease (PD), death due to any cause, discontinuation of treatment for any reason, or initiation of new anticancer therapy. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Time to treatment failure was censored at the date of the last follow-up visit for participants who did not discontinue early, who were still alive, and who have not progressed.
Time Frame: From Date of Randomization to Measured Progressive Disease, Death Due to Any Cause, Discontinuation of Treatment or Initiation of New Anticancer Therapy (Up To 39 Months)
Population: All randomized participants who received at least one dose of study drug during study Phase 2. Censored participants in the GC+N Arm = 1 and in the GC Arm = 0.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 90 | 91
Months | 4.16 [4.01 to 4.24] | 3.75 [2.92 to 4.01]

7. Secondary Outcome: Phase 2: Change From Baseline in EuroQol 5-Dimensional 3 Level (EuroQol-5D-3L) Index Score
Description: EQ-5D measures mobility, self-care, usual activities, pain/discomfort, anxiety/depression. 3 severity levels: no, some, severe problems. The index score was calculated from a set of item weights to derive a score on a theoretical scale of 0 to 1, with 1 representing the best health status and zero representing death based on item weights for the Japanese population. One Cycle = 3 weeks and it can be delayed up to 6 weeks.
Time Frame: Baseline, Cycle 4 (Cycle = 3 weeks)
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post-baseline EQ-5D data during study Phase 2.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 77 | 61
Score on a scale | 0.04 (0.16) | 0.03 (0.17)

8. Secondary Outcome: Phase 2: Change From Baseline in EuroQol 5-Dimensional 3 Level (EuroQol-5D-3L) Visual Analog Scale (VAS)
Description: EQ-5D VAS allowed participants to rate their present health condition. Possible scores ranged from 0 (worst imaginable health state) to 100 (best imaginable health state). One Cycle = 3 weeks and it can be delayed up to 6 weeks.
Time Frame: Baseline, Cycle 4 (Cycle = 3 weeks)
Population: All randomized participants who received at least one dose of study drug and had had evaluable baseline and post-baseline EQ-5D data during study Phase 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 77 | 61
units on a scale | 7.81 (18.90) | 11.10 (18.03)

9. Secondary Outcome: Phase 2: Change From Baseline in Lung Cancer Symptom Scale (LCSS)
Description: The LCSS is a validated and reliable instrument to assess lung cancer-specific symptoms and their impact on QOL.The LCSS total score was defined as the mean of the 9 items of the scale and the average symptom burden index (ASBI) is defined as the mean of 6 symptom-specific lung cancer questions. Each of the 9 symptom or summary items is assessed on a 100-mm visual analogue scale (VAS), with 0 representing no symptoms or better QOL.
Time Frame: Baseline, Cycle 4 (Cycle = 3 weeks)
Population: All randomized participants who received at least one dose of study drug had evaluable baseline and post-baseline LCSS data. One Cycle = 3 weeks and it can be delayed up to 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
Number analyzed (Participants) | 90 | 91
units on a scale
  Loss of Appetite: number analyzed (Participants) | 77 | 61
  Loss of Appetite | -4.48 (26.20) | -9.03 (29.32)
  Fatigue: number analyzed (Participants) | 77 | 61
  Fatigue | -5.42 (26.63) | -4.02 (26.47)
  Cough: number analyzed (Participants) | 77 | 61
  Cough | -18.00 (24.17) | -15.82 (30.59)
  Dyspnea: number analyzed (Participants) | 77 | 61
  Dyspnea | -5.14 (22.51) | -5.08 (24.51)
  Hemoptysis: number analyzed (Participants) | 77 | 61
  Hemoptysis | -4.75 (21.75) | -4.10 (16.46)
  Pain: number analyzed (Participants) | 77 | 61
  Pain | -10.68 (22.07) | -12.38 (26.99)
  Overall Symptoms: number analyzed (Participants) | 77 | 61
  Overall Symptoms | -11.62 (23.20) | -9.56 (24.61)
  Interference: number analyzed (Participants) | 77 | 61
  Interference | -6.92 (26.70) | -5.93 (29.78)
  Quality of Life: number analyzed (Participants) | 77 | 61
  Quality of Life | -5.10 (23.83) | -15.43 (28.46)
  Average Symptom Burden Index (ASBI): number analyzed (Participants) | 77 | 61
  Average Symptom Burden Index (ASBI) | -8.08 (12.81) | -8.40 (16.24)
  LCSS Total Score: number analyzed (Participants) | 77 | 61
  LCSS Total Score | -8.01 (13.64) | -9.04 (16.32)

10. Secondary Outcome: Phase 1b: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Necitumumab
Description: The Cmax is observed maximum serum concentration, taken directly from the serum concentration-time profile.
Time Frame: Cycle 1 (C1) Day 1 (D1) and C3 D1: Predose, End-of-infusion and 1, 3, 6, 24, 96, 168 h post-end-of-infusion
Population: All enrolled participants who had adequate data to calculate at least 1 PK parameter during study Phase 1b. In cohort 1 (cycle 3), zero participants were analyzed because no data was collected for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/ml)
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
micrograms/milliliter (µg/ml)
  Cycle 1 | 454 (6) | 371 (32)
  Cycle 3: number analyzed (Participants) | 0 | 3
  Cycle 3 |  | 372 (15)

11. Secondary Outcome: Phase 1b: PK: Cmax of Gemcitabine and Cisplatin
Description: The Cmax is observed maximum plasma concentration, taken directly from the plasma concentration-time profile.
Time Frame: Gemcitabine: Cycle 1(C1) Day1(D1): Predose, End-of-infusion and 0.5, 1, 2 h post-end-of-infusion; Cisplatin:C1 D1: Predose, End-of-infusion and 3, 21, 93, 165 h post-end-of-infusion
Population: All enrolled participants who had adequate data to calculate at least 1 PK parameter during study Phase 1b.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
nanogram per milliliter (ng/mL)
  Gemcitabine | 17400 (8) | 26000 (16)
  Cisplatin | 3740 (14) | 3980 (10)

12. Secondary Outcome: Phase 1b: PK: Area Under the Serum Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Necitumumab
Description: The AUC(0-infinity) is area under the serum concentration-time curve from time zero to infinite time.
Time Frame: Cycle 1 (C1) Day 1 (D1) and C3 D1: Predose, End-of-infusion and 1, 3, 6, 24, 96, 168 h post-end-of-infusion
Population: All enrolled participants who had adequate data to calculate at least 1 PK parameter during study Phase 1b. In cohort 1 and 2 (cycle 3), zero participants were analyzed because no data was collected for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (µg*h/mL)
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
microgram*hour per milliliter (µg*h/mL)
  Cycle 1: number analyzed (Participants) | 2 | 4
  Cycle 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation not figured due to an N of 2 and the individual minimum-maximum values = 39400-42900. | 38900 (28)
  Cycle 3: number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Phase 1b: PK: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Gemcitabine and Cisplatin
Description: The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time.
Time Frame: Gemcitabine: C1D1: Predose, End-of-infusion and 0.5, 1, 2 h post-end-of-infusion; Cisplatin:C1D1: Predose, End-of-infusion and 3, 21, 93, 165 h post-end-of-infusion
Population: All enrolled participants who had adequate data to calculate at least 1 PK parameter during study Phase 1b. In cohort 1 (cisplatin), zero participants were analyzed because no data was collected for the outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2
Number analyzed (Participants) | 3 | 6
nanogram*hour per milliliter (ng*h/mL)
  Gemcitabine: number analyzed (Participants) | 3 | 4
  Gemcitabine | 8710 (7) | 13300 (19)
  Cisplatin: number analyzed (Participants) | 0 | 1
  Cisplatin |  | NA (NA) — In Cohort 2, summary statistics of t1/2 dependent parameters were not calculated as per the statistical analysis plan because n=1.

14. Secondary Outcome: Phase 2: PK: Minimum Concentration (Ctrough) of Necitumumab
Description: The minimum observed serum concentration (Ctrough) of Necitumumab was evaluated.
Time Frame: Predose Day 1 of Cycle 1, 2, 3, 4, and every 2 cycles after Cycle 5
Population: All enrolled participants who had adequate data to calculate at least 1 PK parameter during study Phase 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab)
Number analyzed (Participants) | 90
microgram per milliliter (µg/mL)
  Dose 3: number analyzed (Participants) | 47
  Dose 3 | 77.9 (30)
  Dose 5: number analyzed (Participants) | 49
  Dose 5 | 110 (32)
  Dose 7: number analyzed (Participants) | 49
  Dose 7 | 130 (36)
  Dose 9: number analyzed (Participants) | 34
  Dose 9 | 137 (41)
  Dose 13: number analyzed (Participants) | 13
  Dose 13 | 145 (48)
  Dose 17: number analyzed (Participants) | 9
  Dose 17 | 120 (59)
  Dose 21: number analyzed (Participants) | 5
  Dose 21 | 194 (44)

15. Secondary Outcome: Phase 2: Number of Participants With Serum Anti-Necitumumab Antibody Assessment (Immunogenicity)
Description: A participant was considered to have an anti-Necitumumab antibody response if anti-drug antibodies (ADA) were detected at any time point.
Time Frame: Baseline up to 30 Days Post Last Infusion (estimated up to 39 months)
Population: All enrolled participants who received at least 1 dose of drug and had evaluable data for antibodies during study Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab)
Number analyzed (Participants) | 90
Participants | 4

ADVERSE EVENTS:
Time Frame: Up To 39 Months
Description: All enrolled participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Phase 1b: Cohort 1: Gemcitabine at a dose of 1000 mg/m^2 (milligrams per square meter) was administered over approximately 30 minutes intravenously (IV) on Days 1 and 8 of each cycle for a maximum of 4 cycles.
- Phase 1b: Cohort 2: Gemcitabine at a dose of 1250 mg/m^2 was administered over approximately 30 minutes IV on Days 1 and 8 of each cycle for a maximum of 4 cycles.
Arm/Group | Phase 1b: Cohort 1 | Phase 1b: Cohort 2 | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) | Phase 2: GC (Gemcitabine, Cisplatin)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 63/90 | 74/91
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 32/90 | 22/91
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 90/90 | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b: Cohort 1 (N=3) | Phase 1b: Cohort 2 (N=6) | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) (N=90) | Phase 2: GC (Gemcitabine, Cisplatin) (N=91)
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 1 (1)
Retroperitoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1b: Cohort 1 (N=3) | Phase 1b: Cohort 2 (N=6) | Phase 2: GC+N (Gemcitabine, Cisplatin + Necitumumab) (N=90) | Phase 2: GC (Gemcitabine, Cisplatin) (N=91)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (8) | 43 (55) | 53 (65)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6) | 3 (3)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (3) | 4 (10) | 5 (10) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 3 (8) | 13 (19) | 13 (25)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4) | 4 (4) | 2 (2) | 7 (9)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 3 (3) | 7 (8)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic nerve disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (7) | 2 (2)
Anal erosion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (5) | 58 (76) | 53 (74)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 26 (43) | 21 (23)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (7) | 5 (10) | 55 (111) | 54 (95)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 3 (5) | 37 (48) | 11 (11)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (5) | 17 (28) | 16 (22)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extravasation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 4 (7) | 6 (7)
Fatigue (General disorders) | 1 (1) | 3 (4) | 17 (39) | 13 (18)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (5)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 4 (7) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 2 (2) | 34 (49) | 32 (44)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 10 (16) | 10 (12)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 18 (18) | 15 (21)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (2) | 7 (9) | 1 (1)
Dacryocanaliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (8) | 5 (5)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 4 (4)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 2 (3) | 44 (48) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea manuum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 11 (12) | 10 (11)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 3 (6)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (4) | 18 (28) | 16 (22)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 17 (27) | 9 (15)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (3) | 9 (10) | 2 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
Blood creatine phosphokinase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 8 (12) | 10 (15)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram st segment depression (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 7 (8) | 3 (3)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 4 (11) | 7 (15)
Neutrophil count decreased (Investigations) | 1 (2) | 3 (7) | 53 (119) | 45 (91)
Platelet count decreased (Investigations) | 1 (1) | 2 (5) | 49 (96) | 46 (81)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 13 (16) | 11 (13)
Weight increased (Investigations) | 0 (0) | 0 (0) | 7 (12) | 5 (8)
White blood cell count decreased (Investigations) | 1 (2) | 2 (2) | 49 (99) | 39 (70)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (6) | 4 (9) | 62 (112) | 48 (87)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 4 (5) | 4 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (6)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 6 (9) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 8 (23) | 11 (19)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 12 (14) | 8 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (5) | 9 (15) | 3 (4)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7) | 35 (54) | 8 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 12 (15) | 24 (36)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5) | 4 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 4 (4)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 6 (6) | 9 (9)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dementia with lewy bodies (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2) | 19 (22) | 9 (11)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 7 (7) | 6 (7)
Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paralysis recurrent laryngeal nerve (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 15 (17) | 19 (24)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 5 (5) | 1 (1)
Haemoglobinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 7 (8) | 5 (6)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0/5 (0) | 0/79 (0) | 1/81 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 0/5 (0) | 1/79 (1) | 0/81 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 12 (12) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (5) | 42 (68) | 49 (86)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 18 (18) | 18 (18)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 72 (79) | 6 (6)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 48 (49) | 8 (8)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 8 (9) | 3 (3)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 10 (11) | 7 (10)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 6 (8) | 11 (12)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
Dermabrasion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 5 (5) | 9 (10)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 2 (5) | 3 (7) | 3 (6)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 4 (6) | 7 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-06-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT01763788/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT01763788/SAP_001.pdf